CLINICAL TRIAL: NCT05783063
Title: Effects of Intermittent Theta Burst Stimulation (iTBS) on Increased Appetite Induced by Antipsychotics in Patients With Schizophrenia
Brief Title: iTBS for Increased Appetite Induced by Antipsychotics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Deputy Director of the Department of Psychiatry, the Second Xiangya Hospital of Central South University., Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WU20221015
Record Dates: First submitted 2023-02-28; First posted 2023-03-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; appetite; weight; antipsychotics; iTBS
MeSH Terms: conditions — Schizophrenia; Body Weight

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial testing iTBS versus sham
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active stimulation (Active Comparator): Intermittent theta burst stimulation to the dorsolateral prefrontal cortex; 5 sessions per day, for 5 days.
  Interventions: Device: Active iTBS
- Sham stimulation (Sham Comparator): Sham stimulation to the dorsolateral prefrontal cortex; 5 sessions per day, for 5 days.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: Active iTBS — Mag-TD
  Arms: active stimulation
Device: Sham iTBS — Mag-TD
  Arms: Sham stimulation

SUMMARY:
Antipsychotics are prone to cause metabolic side effects, including weight gain, hyperglycemia, insulin resistance, hyperlipidemia and so on, leading to a 2-3 times higher risk of death in patients with schizophrenia compared to healthy people. Conventional high-frequency rTMS have been used to treat people with obesity and showed certain effectiveness. However, studies involving schizophrenia patients and intermittent theta burst (iTBS) mode are rarely seen. The goal of this clinical trial is to evaluate the efficacy and safety of iTBS on ameliorating increased appetite induced by antipsychotics in people with schizophrenia.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of iTBS on ameliorating increased appetite induced by antipsychotics in people with schizophrenia by measuring changes in clinical ratings at baseline, after all the treatments, and 2 weeks, 4 weeks after intervention. 60 schizophrenia patients will be randomized to receive active or sham interventions administered to the left dorsolateral prefrontal cortex. The experimental group will be applied to active iTBS rTMS involving 600 pulses (3 minutes), 5x daily at 60 minutes intervals for 5 days. Changes in appetite from baseline to the end of the study will be measured by Three Factor Eating Questionnaire (TFEQ), Food Cravings Questionnaire-Trait (FCQ-T), Food Cravings Questionnaire-State (FCQ-S) and Visual Analogue Scale (VAS). Clinical symptoms and mood status will be assessed by Positive and Negative Symptom Scale (PANSS), the Calgary Depression Scale for Schizophrenia (CDSS) and Clinical Global Impression (CGI). Improvement of cognition could be measured by Delay Discounting Task (DDT), Stop-signal task (SST) and MATRICS (Measurement and Treatment Research to Improve Cognition in Schizophrenia) Consensus Cognitive Battery (MCCB). Changes of appetite related Indicators of glycolipid metabolism and neuroregulatory factor, along with microflora before and after intervention will be recorded by collecting blood and feces specimens. The adverse effect will be evaluated by Treatment Emergent Symptom Scale (TESS) and Adverse Event Record Form (AERF). Task-based magnetic resonance imaging (MRI) and arterial spin labeling (ASL) will be used to measure changes of brain activity associated with food stimuli and cerebral blood flow(CBF) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-40 years old;
2. Meeting the diagnostic criteria for schizophrenia in DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition);
3. BMI ≥ 25kg/m 2 or over 10% weight gain after taking antipsychotics in the last year;
4. Not receiving TMS therapy in the past month;
5. Using no more than two antipsychotic medications (including olanzapine, haloperidol, amisulpride, asenapine, risperidone, paliperidone, clozapine, quetiapine, iloperidone, chlorpromazine, sertindole, zotepine), not using antidepressants, mood stabilizers and other drugs, but allowing short-term use of benzodiazepines, benzhexol and propranolol;
6. Signing written informed consents voluntarily.

Exclusion Criteria:

1. Other severe mental illnesses, mental retardation, dementia and severe cognitive impairment according to diagnostic criteria of ICD-10 or DSM-5;
2. Abnormal brain structure or function owing to any major physical disease, neurological disease, traumatic brain injury, etc.;
3. Metallic implants, pacemakers, epilepsy history or other contraindications of TMS;
4. Suicidal thoughts or behaviors;
5. Alcohol or substance abuse;
6. Pregnant or lactating women;
7. Other contraindications of MRI;
8. Receiving regular MECT, or weight-loss therapy in the latest month;
9. Other abnormal examination results considered to be inappropriate for inclusion by researchers.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in body mass index (BMI) | Baseline, after 5 treatment days, 2 weeks and 4 weeks post-treatment
  Weight gain will be assessed by BMI, caculated by weight in kilograms divided by height in meters squared

SECONDARY OUTCOMES:
Changes in Positive and Negative Symptom Scale (PANSS) | Baseline and 4 weeks post-treatment
  Range from 30 to 210, higher score indicates more severe positive and negative symptoms.
Changes in Calgary Depression Scale for Schizophrenia (CDSS) | Baseline and 4 weeks post-treatment
  Range from 0 to 27, higher score indicates more severe affective symptoms.
Changes in the Clinical Global Impressions (CGI) | Baseline and 4 weeks post-treatment
  The Clinical Global Impressions (CGI) scale, quantifying the severity of psychopathology, ranging from 1 to 7 and improvements, ranging from 1 to 7 after treatments
Changes in brain perfusion. | Baseline, after 5 treatment days and 4 weeks post-treatment
  The arterial spin labeling (ASL) pulse sequences to quantify the cerebral blood flow (CBF).
Changes in brain function. | Baseline, after 5 treatment days and 4 weeks post-treatment
  Functional MRI (fMRI) based on the blood oxygen level dependent (BOLD) contrast that can detect changes in blood oxygenation to analyze the change of brain function after intervention.
Changes in MCCB | Baseline and 4 weeks post-treatment
  The MATRICS™ Consensus Cognitive Battery
Changes in SST. | Baseline, after 5 treatment days, 2 weeks and 4 weeks post-treatment
  Stop-signal task (SST) will be used to assess cognitive control.
Changes in DDT. | Baseline, after 5 treatment days, 2 weeks and 4 weeks post-treatment
  Delay Discounting Task (DDT) will be used to assess impulsiveness in decision making.
Changes in the Three-factor Eating Questionnaire (TFEQ) | Baseline, after 5 treatment days, 2 weeks and 4 weeks post-treatment
  TFEQ includes three domains, cognitive restraint, uncontrolled eating and emotional eating, range from 21 to 84, higher scores indicates higher appetite.
Changes in the Food Cravings Questionnaire-Trait (FCQ-T) | Baseline, after 5 treatment days, 2 weeks and 4 weeks post-treatment
  Food Cravings Questionnaire-Trait (FCQ-T) is a six-point Likert scale to measure individuals' stable food craving traits containing nine factors with 39 items.
Changes in the Food Cravings Questionnaire-State (FCQ-S) | Baseline, after 5 treatment days, 2 weeks and 4 weeks post-treatment
  The Food Cravings Questionnaire-State (FCQ-S) is a five-point Likert scale that measures the intensity of momentary food craving.
Changes in the visual analogue scale (VAS) | Everyday from baseline to 4 weeks after treatment
  The visual analogue scale (VAS) will be used to assess the subjective sense of appetite covering hungry, satiety, desire to eat, and overeating, scoring from 0 = "not at all" to 10 = "extremely".
Changes in the types of intestinal flora. | Baseline and 4 weeks post-treatment
  Feces will be collected and DNA will be extraced for quantitative analysis of intestinal flora composition.
Changes in plasma agouti related regulatory proteins. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in ng/mL.
Changes in plasma serum proopioid-melanocortin. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in ng/mL.
Changes in plasma serum ghrelin. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in ng/mL
Changes in plasma serum leptin. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in ng/mL.
Changes in the proportion of of intestinal flora. | Baseline and 4 weeks post-treatment
  Feces will be collected and DNA will be extraced for quantitative analysis of intestinal flora composition.
Changes in plasma prolactin. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mcg/L.
Changes in serum total bile acids. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mmol/l.
Changes in glycosylated hemoglobin. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mmol/mol.
Changes in serum Low-density lipoprotein cholesterol. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mg/dl.
Changes in serum high-density lipoprotein cholesterol. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mg/dl.
Changes in serum total cholesterol. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mg/dl.
Changes in serum triglycerides. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mmol/l.
Changes in serum glucagon-like peptide-1. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in pmol/l.
Changes in serum glucagon. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in ng/l.
Changes in serum fasting insulin. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mmol/l.
Changes in serum fasting blood glucose. | Baseline, after 5 treatment days and 4 weeks post-treatment
  in mmol/l.

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, M.D. Ph.D, Principal Investigator — Department of Psychiatry, The Second Xiangya Hospital of Central South University
Locations (2):
- China (2):
  - Central South University, Changsha, Hunan
  - The Second People's Hospital of Dali Bai Autonomous Prefecture, Dali, Yunnan

IPD SHARING:
Plan to Share IPD: No
Data Sharing Plan The proposed study will involve a small sample (60 patients with schizophrenia) recruited from clinical institutions of the Second People's Hospital of Dali Bai Autonomous Prefecture and the Second Xiangya Hospital of Central South University in China. The final dataset will comprise self-reported demographic and clinical characteristics, behavioral and neuroimaging data, along with laboratory data from blood and stool specimens provided by the participants. Because schizophrenia is a reportable severe mental disorder, identifying information will be collected. Although the final dataset is deidentified before it is released for sharing, we believe it is still possible to infer the disclosure of subjects with psychotic characteristics. Patients with schizophrenia belong to a vulnerable group, often accompanied by a sense of stigma. Given the social distress of the participants and the relatively limited area in which we recruited the participants, we thought it would

REFERENCES:
- [Derived] Qin Y, Yang J, Xu B, Yang J, Chen H, Zou T, Teng Z, Liu J, Zhang T, Su Y, Wu R, Dong Z, Yang C, Huang J. Effects of intermittent theta burst stimulation (iTBS) on appetite change and body weight in inpatients with schizophrenia in China: study protocol for a randomised controlled trial. BMJ Open. 2025 Apr 8;15(4):e090932. doi: 10.1136/bmjopen-2024-090932. PMID 40204331